CLINICAL TRIAL: NCT01987986
Title: A Phase 2, Double-blind and Placebo Dose Ranging Study of Repeat Doses of AA4500 for the Treatment of Edematous Fibrosclerotic Panniculopathy
Brief Title: A Phase 2, Randomized, Double-blind, Placebo Controlled Dose Ranging Study of Repeat Doses of AA4500 for the Treatment of Edematous Fibrosclerotic Panniculopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUX-CC-831
Record Dates: First submitted 2013-10-30; First posted 2013-11-20 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Edematous Fibrosclerotic Panniculopathy (EFP)
Keywords: cellulite; dimple; orange peel; cottage cheese; mattress texture
MeSH Terms: conditions — Cellulite | interventions — Microbial Collagenase; xiapex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AA4500 0.06 mg (low dose) (Experimental): AA4500 (Collagenase Clostridium Histolyticum)
  Each subject could receive up to three treatment sessions. Each treatment session was separated by approximately 21 days.
  Interventions: Biological: Collagenase Clostridium Histolyticum
- AA4500 0.48 mg (mid-dose) (Experimental): AA4500 (Collagenase Clostridium Histolyticum)
  Each subject could receive up to three treatment sessions. Each treatment session was separated by approximately 21 days.
  Interventions: Biological: Collagenase Clostridium Histolyticum
- AA4500 0.84 mg (high dose) (Experimental): AA4500 (Collagenase Clostridium Histolyticum)
  Each subject could receive up to three treatment sessions. Each treatment session was separated by approximately 21 days.
  Interventions: Biological: Collagenase Clostridium Histolyticum
- Placebo (Placebo Comparator): Placebo
  Each subject could receive up to three treatment sessions. Each treatment session was separated by approximately 21 days.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Collagenase Clostridium Histolyticum — injectible intervention
  Other Names: AA4500; Xiaflex; Xiapex
  Arms: AA4500 0.06 mg (low dose); AA4500 0.48 mg (mid-dose); AA4500 0.84 mg (high dose)
Biological: Placebo
  Arms: Placebo

SUMMARY:
To assess the safety and effectiveness of repeat doses of AA4500 in the treatment of edematous fibrosclerotic panniculopathy (EFP) commonly known as cellulite in adult women.

DETAILED DESCRIPTION:
The Phase 2a study is a randomized, double-blind multiple-dose study that is expected to enroll approximately 144 women between the ages of 18 and 45 in the United States. Treatment effectiveness will be evaluated by investigator and patient assessments, as well as 3-D photographic imaging techniques. Once the safety and local tolerability profile from the first stage has been found to be acceptable subjects will be enrolled in stage 2. After an interim safety and local tolerability review was completed of all subjects in stage 1, it was determined that enrollment in stage 2 is acceptable and has been initiated.

ELIGIBILITY:
Inclusion Criteria:

1. Be a female between 18 to 45 years of age.
2. Have at least one well defined dimple that is at least 1 cm but not more than 2 cm along the long axis and that is evident when the subject is standing
3. Have a photonumeric cellulite severity scale (CSS) score between 6 and 12
4. Have a Body Mass Index (BMI) >19 and <30 kg/m2, and intends to maintain stable body weight throughout the duration of the study
5. Be willing to apply appropriate sunscreen to the selected quadrant before each exposure to the sun while participating in the study
6. Be judged to be in good health, based upon the results of a medical history, physical examination, and laboratory profile at screening.
7. Have a negative urine pregnancy test at screening and before injection of AA4500 and be using an effective contraception method (ie, abstinence, intrauterine device [IUD], hormonal [estrogen/progestin] contraceptives, or barrier control) for at least one menstrual cycle prior to study enrollment and for the duration of the study.
8. Be willing and able to cooperate with the requirements of the study.
9. Voluntarily sign and date an informed consent agreement approved by the Institutional Review Board/Independent Ethics Committee/Human Research Ethics Committee (IRB/IEC/HREC).
10. Be able to read, complete and understand the Patient Reported Outcomes rating instruments in English.

Exclusion Criteria:

1. Thyroid disease, unless controlled with medication for ≥ 6 months
2. Uncontrolled diabetes mellitus, as determined by the investigator
3. Uncontrolled hypertension, as determined by the investigator
4. Vascular disorder (eg, phlebitis or varicose veins) in area to be treated
5. Lipedema or a lymphatic disorder
6. Cushing's disease and/or use of systemic corticosteroids
7. History of lower extremity thrombosis or post-thrombosis syndrome
8. Documented autoimmune disorder such as lupus erythematosus, rheumatoid arthritis
9. Inflammation or active infection in area to be treated
10. Cutaneous alteration in area to be treated
11. Rash, eczema, psoriasis, or skin cancer in the area to be treated
12. History of keloidal scarring or abnormal wound healing
13. Coagulation disorder
14. Taking a medication for chronic anticoagulation (except for ≤ 150 mg aspirin daily)
15. Known active hepatitis A, B or C
16. Known immune deficiency disease or a positive test for human immunodeficiency virus (HIV)
17. Other significant conditions including body dysmorphic disorder, which in the investigator's opinion would make the subject unsuitable for enrollment in the study
18. Is menopausal defined as 12 months of amenorrhea in the absence of other biological or physiological causes, as determined by the investigator
19. Has used any of the following for the treatment of EFP on the legs or buttock within the timelines identified below or intends to use any of the following at any time during the course of the study:

    * Liposuction on the side of the body selected for treatment during the 12-month period before injection of AA4500
    * Injections (eg, mesotherapy); radiofrequency device treatments; laser treatment; or surgery (including subcision) within the selected treatment quadrant during the 12-month period before injection of AA4500
    * Endermologie or similar treatments within the selected treatment quadrant during the 6-months period before injection of AA4500
    * Massage therapy within the selected treatment quadrant during the 3-month period before injection of AA4500
    * Creams (eg, Celluvera™, TriLastin®) to prevent or mitigate EFP within the selected treatment quadrant during the 2-week period before injection of AA4500
20. Has a tattoo located within 2 cm of the site of injection
21. Is presently nursing a baby or providing breast milk for a baby.
22. Intends to become pregnant during the study.
23. Intends to initiate an intensive sport or exercise program during the study.
24. Has received an investigational drug or treatment within 30 days before injection of AA4500.
25. Has a known systemic allergy to collagenase or any other excipient of AA4500.
26. Has received any collagenase treatments within 30 days before treatment.

    -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Urdaneta, MD MPH, Study Director — Endo Pharmaceuticals
Locations (10):
- United States (10):
  - Dermatology Cosmetic Laser Medical Associates of La Jolla, San Diego, California
  - ATS Clinical Research, Santa Monica, California
  - Dermatology Research Institute, Coral Gables, Florida
  - Kenneth Beer, MD PA, West Palm Beach, Florida
  - Mercy Health Research, Washington, Missouri
  - Sadick Research Group, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Charlottesville Dermatology, Charlottesville, Virginia
  - Premier Clinical Research, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- AA4500 0.06 mg (Low Dose); AA4500 0.48 mg (Mid-dose); AA4500 0.84 mg (High Dose): AA4500 (Collagenase Clostridium Histolyticum)
  Each subject could receive up to three treatment sessions. Each treatment session was separated by approximately 21 days.
  Collagenase Clostridium Histolyticum: injectible intervention
- Placebo: Placebo
  Each subject could receive up to three treatment sessions. Each treatment session was separated by approximately 21 days.
  Placebo
Period: Overall Study
Arm/Group | AA4500 0.06 mg (Low Dose) | AA4500 0.48 mg (Mid-dose) | AA4500 0.84 mg (High Dose) | Placebo
Started | 43 | 43 | 40 | 24
Completed | 41 | 43 | 38 | 24
Not Completed | 2 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AA4500 0.06 mg (Low Dose) | AA4500 0.48 mg (Mid-dose) | AA4500 0.84 mg (High Dose) | Placebo | Total
Number analyzed (Participants) | 43 | 43 | 40 | 24 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (5.78) | 36.8 (7.07) | 36.1 (5.62) | 37.3 (8.08) | 36.9 (6.50)
Age, Customized [Count of Participants; unit: Participants]
  <25 | 2 | 3 | 2 | 1 | 8
  25-34 | 6 | 11 | 12 | 6 | 35
  35-44 | 33 | 23 | 25 | 13 | 94
  >=45 | 2 | 6 | 1 | 4 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 40 | 24 | 150
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 13 | 9 | 4 | 36
  Not Hispanic or Latino | 33 | 30 | 31 | 20 | 114
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 1 | 1
  Black or African American | 2 | 3 | 4 | 2 | 11
  White | 40 | 40 | 36 | 20 | 136
  Other | 1 | 0 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 43 | 43 | 40 | 24 | 150

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment of Aesthetic Improvement
Description: Investigators assessment of aesthetic improvement (I-GAIS) scores ranged from 3 to -1 as follows: 3 (very much improved), 2 (much improved), 1 (improved), 0 (no change), -1 (worse).
Time Frame: Baseline, Day 73
Population: All subjects who received at least one injection of study drug and had at least one post-injection efficacy measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 0.06 mg (Low Dose) | AA4500 0.48 mg (Mid-dose) | AA4500 0.84 mg (High Dose) | Placebo
Number analyzed (Participants) | 43 | 43 | 40 | 24
units on a scale | 0.7 (0.82) | 0.9 (0.93) | 1.1 (0.91) | 0.5 (0.72)

2. Other Pre Specified Outcome: Investigator Cellulite Severity Score (CSS) Total Score- Change From Baseline
Description: The CSS is a photonumeric scale that was used to evaluate 5 morphologic features of cellulite; (A) number of evident depressions, (B) depth of depressions, (C) morphological appearance of skin surface alterations, (D) laxity, flaccidity or sagging of skin, and (E) current classification scale based on medical literature including Nuernberger and Mueller. The severity of each feature is rated on a scale from 0 (none) to 3 (most severe). The CSS total score is the sum of the 5 cellulite features (range: 0 to 15, with higher scores corresponding to more severe cellulite). Change is Day 73 study visit rating minus baseline rating; negative values indicate improvement in cellulite.
Time Frame: Baseline, Day 73
Population: All subjects who received at least one injection of study drug and had at least one post-injection efficacy measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 0.06 mg (Low Dose) | AA4500 0.48 mg (Mid-dose) | AA4500 0.84 mg (High Dose) | Placebo
Number analyzed (Participants) | 43 | 43 | 40 | 24
units on a scale | -1.1 (1.74) | -1.3 (1.70) | -1.9 (2.37) | -0.7 (1.52)

3. Other Pre Specified Outcome: Subject Cellulite Severity Item (CSI)-Change From Baseline
Description: CSI scores ranged from 0 (no cellulite present), 1 (very mild), 2 (mild), 3 (moderate), 4 (severe) to 5 (very severe). Change is Day 73 study visit rating minus baseline rating; negative values indicate a lessening in cellulite severity.
Time Frame: Baseline, Day 73
Population: All subjects who received at least one injection of study drug and had at least one post-injection efficacy measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 0.06 mg (Low Dose) | AA4500 0.48 mg (Mid-dose) | AA4500 0.84 mg (High Dose) | Placebo
Number analyzed (Participants) | 43 | 43 | 40 | 24
units on a scale | -0.7 (1.22) | -1.1 (1.07) | -1.3 (1.34) | -0.8 (1.35)

4. Other Pre Specified Outcome: Subject Global Bother Assessment (SGBA)- Change From Baseline
Description: Subjects rated their cellulite on a scale from 0 (not at all bothered) to 4 (extremely bothered). Change from baseline is Day 73 study visit value minus baseline value; negative change reflects an improvement in the amount the subject was bothered by cellulite; positive change reflects a worsening in the amount the subject is bothered by cellulite.
Time Frame: Baseline, Day 73
Population: All subjects who received at least one injection of study drug and had at least one post-injection efficacy measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 0.06 mg (Low Dose) | AA4500 0.48 mg (Mid-dose) | AA4500 0.84 mg (High Dose) | Placebo
Number analyzed (Participants) | 43 | 43 | 40 | 24
units on a scale | -0.9 (1.33) | -1.0 (1.23) | -1.0 (1.12) | -1.0 (1.33)

5. Other Pre Specified Outcome: Subject-reported Cellulite Impact Scale (SR-CIS)-Change From Baseline
Description: Subjects were asked to answer 6 exploratory questions regarding the appearance of their cellulite on a scale of 0 to 10 with 0 representing "not at all" and 10 representing "extremely." A SR-CIS total score was derived from these 6 questions with values varying from 0 (No negative impact) to 60 (Extreme negative impact). Change from baseline is Day 73 value minus baseline value; negative change reflects an improvement.
Time Frame: Baseline, Day 73
Population: All subjects who received at least one injection and who had at least one post-injection efficacy measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 0.06 mg (Low Dose) | AA4500 0.48 mg (Mid-dose) | AA4500 0.84 mg (High Dose) | Placebo
Number analyzed (Participants) | 43 | 43 | 40 | 24
units on a scale | -15.0 (18.9) | -18.0 (15.70) | -17.7 (14.61) | -11.9 (13.97)

6. Other Pre Specified Outcome: Subject Satisfaction With Treatment Assessment (SCTA)
Description: Subjects rated their treatment satisfaction at the Day 73 visit on a 5-point scale ranging from -2 (very dissatisfied) to +2 (very satisfied)
Time Frame: Day 73
Population: All subjects who received at least one injection of study drug and had at least one post -injection efficacy measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 0.06 mg (Low Dose) | AA4500 0.48 mg (Mid-dose) | AA4500 0.84 mg (High Dose) | Placebo
Number analyzed (Participants) | 43 | 43 | 40 | 24
units on a scale | 0.0 (1.31) | 0.9 (0.89) | 0.7 (0.93) | 0.1 (1.33)

7. Other Pre Specified Outcome: Subject Global Assessment Cellulite (SGA-C)
Description: Subjects assessed their cellulite based on a 5-point scale from -1 (slightly worse), 0 (same), 1 (slightly improved), 2 (moderately improved), to 3 (much improved) on Day 73
Time Frame: Day 73
Population: All subjects who at least one injection of study drug and had at least one post-injection efficacy measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 0.06 mg (Low Dose) | AA4500 0.48 mg (Mid-dose) | AA4500 0.84 mg (High Dose) | Placebo
Number analyzed (Participants) | 43 | 43 | 40 | 24
units on a scale | 0.9 (1.23) | 1.6 (0.85) | 1.5 (1.04) | 0.8 (0.96)

8. Other Pre Specified Outcome: Subject Global Assessment of Aesthetic Improvement (C-GAIS)
Description: Subjects's assessment of aesthetic improvement (C-GAIS) scores ranged from 3 to -1 as follows: 3 (very much improved), 2 (much improved), 1 (improved), 0 (no change), -1 (worse).
Time Frame: Day 73
Population: All subjects who received at least one injection of study medication and had at least one post injection efficacy measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500 0.06 mg (Low Dose) | AA4500 0.48 mg (Mid-dose) | AA4500 0.84 mg (High Dose) | Placebo
Number analyzed (Participants) | 43 | 43 | 40 | 24
units on a scale | 0.9 (1.14) | 1.6 (0.88) | 1.4 (1.03) | 0.7 (0.91)

ADVERSE EVENTS:
Arm/Group | AA4500 0.06 mg (Low Dose) | AA4500 0.48 mg (Mid-dose) | AA4500 0.84 mg (High Dose) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43 | 0/40 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/43 | 0/43 | 0/40 | 0/24
Other Adverse Events (participants affected / at risk) | 28/43 | 31/43 | 31/40 | 7/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AA4500 0.06 mg (Low Dose) (N=43) | AA4500 0.48 mg (Mid-dose) (N=43) | AA4500 0.84 mg (High Dose) (N=40) | Placebo (N=24)
Pharyngeal absess (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 0.06 mg (Low Dose) (N=43) | AA4500 0.48 mg (Mid-dose) (N=43) | AA4500 0.84 mg (High Dose) (N=40) | Placebo (N=24)
Injection site brusing (General disorders) | 27 (51) | 30 (60) | 28 (58) | 6 (7)
Injection site pain (General disorders) | 11 (15) | 18 (38) | 21 (41) | 2 (4)
Injection site pruritus (General disorders) | 0 (0) | 5 (8) | 7 (10) | 0 (0)
Injection site swelling (General disorders) | 3 (3) | 7 (14) | 5 (8) | 0 (0)
Injection site discoloration (General disorders) | 0 (0) | 5 (6) | 6 (6) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other